CLINICAL TRIAL: NCT03443908
Title: Early Diagnosis and Treatment of Sleep Disordered Breathing in Lung Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped due to lack of enrollment.
Sponsor: Mark M. Fuster, MD (Other)
Responsible Party: Sponsor-Investigator, Mark M. Fuster, MD, Associate Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 161552
Record Dates: First submitted 2018-02-01; First posted 2018-02-23 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Lung Cancer
Keywords: lung cancer; non small cell lung cancer; nsclc; small cell lung cancer; sclc; metastic lung mass; sleep disordered breathing; sdb; obstructive sleep apnea
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CPAP therapy: CPAP therapy (minimum of 3-4 weeks)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP therapy 3-4 weeks
  Other Names: continuous positive airway pressure

SUMMARY:
Sleep-disordered breathing at night is a common medical problem. It leads to daytime fatigue, impairment in concentration and daily activities, and a higher risk of cardiovascular disease and life-threatening events. A particularly common form is obstructive sleep apnea (OSA), and it is usually treatable with a high rate of patient satisfaction and improved quality of life using a continuous positive airway pressure (CPAP) device.

Treatment of this condition improves nighttime low-oxygen levels by ensuring patency of the upper airways. Research shows that in cancer, sleep disordered breathing is frequent. Low oxygen levels overnight may cause tumors to grow: tumors deprived of oxygen grow more blood vessels to try to get more oxygen, and growing more blood vessels makes the tumor grow. This study aims to examine how treating sleep-disordered breathing may lessen blood-flow to lung tumors, and thus serve to ultimately block tumor growth.

Participants of this study will undergo sleep study and receive CPAP therapy as a part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung cancer in one of 2 sub-types:

  1. newly diagnosed early-stage tumor
  2. advanced-stage lung tumor undergoing serial contrast-CT imaging according to standard of care
* Diagnosis of a metastatic carcinomatous mass in the lung
* Positive study for sleep-disordered breathing (SDB) with intermittent hypoxia (IH) and clinical recommendation for CPAP
* Ability and willingness to undergo baseline and repeat perfusion-CT imaging following 3- to 4 weeks of CPAP therapy for SDB (regardless of CPAP compliance).

Note: Participants will undergo sleep study and receive CPAP therapy as a part of routine care.

Exclusion Criteria:

* Lung cancer with a negative sleep study (i.e., no SDB)
* History of radio-contrast allergy
* At excessive risk for contrast nephropathy (following standard radiology renal-risk criteria)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
tumor perfusion | 3-4 weeks
  maximum attenuation value (MAV) detected by perfusion-CT imaging

SECONDARY OUTCOMES:
reduction in circulating tumor cells (CTC) | 3-4 weeks
Reduction in tumor promoting micro RNA expression | 3-4 weeks
Reduction in nocturnal hypoxia | 3-4 weeks
Improvement in sleep quality | 3-4 weeks
progression-free survival (PFS) | 2 years
overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fuster, MD, Principal Investigator — Universityof California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No